CLINICAL TRIAL: NCT00480441
Title: A Phase II Double-Blind Placebo-Controlled Trial of Dronabinol and BRENDA for the Treatment of Cannabis Withdrawal
Brief Title: Effectiveness Study of Dronabinol and BRENDA for the Treatment of Cannabis Withdrawal
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Marina Goldman, Principal Investigator, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5P60DA005186-19 (NIH); 5P60DA005186-19 (NIH)
Record Dates: First submitted 2007-05-30; First posted 2007-05-31 (Estimated); Results first posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Marijuana Dependence
Keywords: Marijuana; Addiction; Substance Withdrawal Syndrome; Clinical Trial; Dronabinol; Behavioral Therapy; Adults; Neuroimaging; Neuropsychological Testing; Neurocognitive Testing; Behavioral Probes
MeSH Terms: conditions — Marijuana Abuse; Behavior, Addictive; Substance Withdrawal Syndrome | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Dronabinol+ BRENDA therapy
  Interventions: Drug: Dronabinol; Behavioral: BRENDA therapy
- 2 (Placebo Comparator): Placebo+BRENDA therapy
  Interventions: Behavioral: BRENDA therapy; Drug: Placebo

INTERVENTIONS:
Drug: Dronabinol — 10mg capsules taken 4 times daily for 2 weeks and then tapered over 1 week
  Other Names: Marinol
  Arms: 1
Behavioral: BRENDA therapy — weekly therapy sessions for 6 weeks
Drug: Placebo — 4 capsules daily for 2 weeks followed by a 1 week taper
  Arms: 2

SUMMARY:
This treatment study is targeted specifically for those who want to stop using marijuana. We want to find out if patients who are dependent on marijuana and want to stop using are helped by a combination of the drug dronabinol and six sessions of individual therapy (BRENDA). Dronabinol is a pill form of the active ingredient in marijuana (THC). Currently, dronabinol is approved for the treatment of nausea in people receiving cancer chemotherapy and as an appetite stimulant in people with AIDS.

In some studies, dronabinol reduced the amount of psychological and physical discomfort experienced when people stopped using marijuana. One purpose of our study is to see if people who are on dronabinol have fewer problems with psychological and physical discomfort than those who are on a placebo.

In addition to treatment, this research trial will also be measuring the reactions of subjects to drug-related cues, and also to computer-presented tasks unrelated to drug use. We may examine whether the response to these cues/tasks either predicts treatment outcome, or is affected by your treatment. This information may also help us to understand the ways in which chronic drug use causes changes in our subjects' mental functioning and how those changes respond to treatment.

In addition to participation in the treatment research trial, some subjects may be asked to undergo a brain scan in an MRI. The purpose of the brain scan research project is to measure brain reactions with a non-invasive, non-radioactive imaging technique known as fMRI (functional magnetic resonance imaging) in marijuana subjects before and after treatment with the medication dronabinol or with an inactive substance (placebo).

DETAILED DESCRIPTION:
1. Background: Cannabis is the most widely used illicit drug in the U.S. According to the 2004 U.S. The 2004 NSDUH estimates there are 3.2 million daily or almost daily marijuana smokers in the United States. Recent reports have estimated that 1.5% of the US population meets DSM-IV diagnostic criteria for cannabis abuse or dependence, with the sharpest increases among young black men and women and young Hispanic men (2). Cannabis users commonly endorse adverse psychosocial and medical effects from their cannabis use, which include dysphoria, loss of control over use, cognitive impairment, and strained social relationships.

In humans, the cannabis withdrawal syndrome is a constellation of affective and behavioral symptoms that occur within 24 to 48 hours after abrupt cessation of marijuana use with a gradual return to baseline after 1-2 weeks. A recent review of the literature on cannabis withdrawal identified consistent reports of anxiety, irritability, physical discomfort, insomnia, and appetite suppression to be associated with abrupt cessation of cannabis use in heavy users across controlled inpatient and outpatient trials.

The agonist dronabinol (Marinol) has shown promise in the prevention of cannabis withdrawal in human lab studies and its reported amelioration of anxiety, misery, insomnia, drug craving and appetite suppression from abrupt cannabis cessation provides the rationale for its use as an agent to prevent cannabis withdrawal in an outpatient, treatment seeking population(9). Dronabinol has also been used as a brief "maintenance" treatment in a cannabis self-administration study in humans. Currently, dronabinol is indicated for treatment of AIDS-related anorexia and nausea associated with cancer chemotherapy. Two principle aims of our proposal are therefore to gain familiarity with cannabis withdrawal in a naturalistic outpatient treatment setting and compare an agonist therapy to placebo to attenuate cannabis withdrawal and enhance treatment outcome.

The general pattern of low rates of total abstinence and lack of significant differences between high intensity psychotherapy treatment vs. low intensity and voucher-based treatment holds across all psychosocial treatment studies. In keeping with prior evidence supporting the relative efficacy of brief interventions for cannabis dependence, the current proposal will apply a well-established brief medicalized psychotherapy known as B.R.E.N.D.A. for the treatment of cannabis dependence.

To date, studies evaluating cannabis patients have primarily focused on identifying neurotoxic drug effects such as impaired learning, memory, attention and executive function. We propose to more fully examine the behaviors with relevance to addiction vulnerability and relapse. Such behaviors include but are not limited to poor inhibition, high risk-taking, positive affective bias toward drug stimuli, poor affect regulation, and poor decision-making. We plan to utilize standardized tasks and questionnaires to objectively characterize dimensions of these addiction relevant behaviors in cannabis patients and to examine the effect of cannabis withdrawal and dronabinol treatment on these behavioral measures. We will also correlate brain differences (structural and functional) with behavioral measures in cannabis dependent patients before and after treatment with dronabinol as compared to placebo.

The search for effective treatment of addictive disorders is limited by our incomplete knowledge about the brain substrates critical for addiction and for addiction recovery. The recent use of PET and fMRI has allowed researchers to examine connections between brain activity and vulnerability to addiction and relapse. In marijuana users, PET and fMRI techniques have been used to study regional brain volumes, blood flow, metabolism. However, understanding cue induced craving is more immediately relevant to treatment and relapse prevention in cannabis addiction since cannabis users have a high rate of relapse compared to those found for other drugs of abuse. In addiction, cues that have been consistently associated with drug reward can trigger craving for the drug. Clinically, the craving for the drug is sufficiently compelling in many cases to precipitate a relapse despite significant effort on the patient's part to maintain abstinence and despite significant negative consequences. Although PET and fMRI techniques have been successfully used to study cue induced craving in other drugs of abuse (e.g. cocaine) leading to greater understanding of the mechanism of relapse (limbic activation in response to drug cues), these techniques have not been utilized in cannabis patients. Several preliminary studies used patient self-report to demonstrate cue induced craving in cannabis patients. We propose to utilize physiological measures and functional neuroimaging to objectively demonstrate cue-induced craving in cannabis dependent subjects and to identify the brain substrates that mediate this craving. Similarly, dronabinol reduced self-reported drug craving in one recent human laboratory study. We propose to examine whether dronabinol will change physiological measures and brain activation in response to drug cues.

2. Study objectives:

1. To evaluate the cannabis withdrawal syndrome in a naturalistic outpatient setting as one possible cause for the low rates of total abstinence seen in our trial and all other clinical trials of adult cannabis dependence.

   1. Primary Hypothesis: Subjective ratings of cannabis withdrawal can be assessed reliably in an outpatient treatment setting.
   2. Secondary Hypothesis: Subjects with high subjective ratings of cannabis withdrawal will have lower rates of abstinence regardless of treatment group (dronabinol vs. placebo).
2. To determine the feasibility and efficacy of a three-week trial of a cannabinoid agonist medication under double blind placebo controlled conditions to treat cannabis withdrawal.

   1. Primary Hypothesis: Dronabinol can be used safely at a dosage of 10mg qid (four times per day) as an outpatient treatment for cannabis withdrawal
   2. Secondary Hypothesis: Dronabinol will perform better than placebo in attenuating the symptoms of cannabis withdrawal.
3. To determine the feasibility and efficacy of providing brief psychotherapy (BRENDA) to patients seeking treatment for cannabis dependence.

   1. Primary Hypothesis: Six sessions of BRENDA therapy can be applied to the treatment of cannabis dependence.
   2. Secondary Hypothesis: Six-sessions of BRENDA therapy for cannabis dependence is an adequate "dose" of individual therapy for subjects motivated to stop smoking marijuana.
4. To characterize the neurocognitive aspects (e.g. attention, working memory, impulsivity, decision making, risk-taking, affective bias/drug preference, reward and punishment sensitivity, affect regulation) of cannabis dependence, cannabis withdrawal and dronabinol effects by utilizing a battery of tasks, questionnaires and interviews.

   1. Primary Hypothesis: Poor performance on neurocognitive tasks and questionnaires will be correlated with duration and amount of cannabis use.
   2. Secondary Hypothesis: Cannabis withdrawal will be correlated with impaired performance on neurocognitive tasks and questionnaires. Dronabinol treatment will reduce this impairment on tasks of affect regulation and affective bias/drug preference compared to placebo.
5. To objectively demonstrate cue-induced craving in cannabis dependent patients and to determine whether baseline measures of our cannabis patients' brain vulnerabilities (of structure, and of function; e.g., resting perfusion) can predict both brain and behavioral outcomes.

   1. Primary Hypothesis: Cue-induced craving will be positively correlated with changes in physiological measures and increased amygdalar activation and negatively correlated with prefrontal activation in cannabis dependent patients during cannabis discontinuation, and dronabinol treatment will reduce the intensity of cue- induced physiological changes and brain activation compared to placebo.
   2. Secondary Hypotheses: Measures of prefrontal cortex gray matter and resting perfusion in prefrontal cortex, cingulate cortex and amygdala will be positively correlated with performance on neurocognitive tasks and questionnaires as well as treatment outcome.

3. Location: This is a single site study. All patient recruitment and data collection will occur at the Treatment Research Center at the University of Pennsylvania, 3900 Chestnut Street, Philadelphia, PA 19104, except for the Neuroimaging which will take place at the HUP6 fMRI in the basement of the Hospital of the University of Pennsylvania, 34th and Spruce Streets, Philadelphia, PA 19104.

STUDY DESIGN

4. Research design & methodology: This is a Phase 2 double blind placebo controlled trial. We will recruit 60 cannabis dependent subjects and treat them with the combination of dronabinol 10mg QID (four times per day) and BRENDA or placebo qid (four times per day) and BRENDA to reduce their consumption of cannabis. Subjects will be 60 men and women with current DSM-IV diagnosis of cannabis dependence. All patients will receive six sessions of BRENDA at visits 1, 3, 6, 9, 11, and 12. The study length for each patient will be one week for screening and baseline self-report and neurocognitive battery measures. Patients who qualify will be offered an opportunity to participate in the fMRI portion of the study with baseline fMRI obtained in the first week prior to starting medications and second fMRI obtained during week two of medications. This is followed by 3 weeks of medication and, after completing medications, three additional weekly visits (two for BRENDA and one for final assessment).

5. Duration: Each subject will participate in a 7 week treatment trial with the following schedule of visits: STUDY VISITS

Week 1 (Baseline Measures):

Week 2 - 4 (Medication Treatment):

Weeks 5-6 (Medication Washout)

Week 7 (Final Visit):

We anticipate that we will require two years to complete data collection with 60 subjects and will require one year for data analysis. Thus, the proposed study will be completed in approximately three years.

SUBJECT SELECTION & WITHDRAWAL

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, 18-55 years old
2. Meets DSM-IV criteria for Cannabis Dependence
3. History of chronic cannabis use of moderate intensity defined by 10 or more years of use with an average frequency of 2 or more joints/day on 5 or more days/week
4. Live within a commutable distance of the Treatment Research Center
5. Understand and sign the informed consent
6. Voluntarily seeking treatment for cannabis dependence

Exclusion Criteria:

1. Current DSM-IV diagnosis of any psychoactive substance dependence other than marijuana, or nicotine dependence
2. Concomitant treatment with sedative hypnotics, opioid analgesics or other known CNS depressants at a dose and frequency that is unacceptable to the principal investigator
3. Mandated to treatment based upon a legal decision or as a condition of employment
4. Current severe psychiatric symptoms, e.g. psychosis, dementia, acute suicidal or homicidal ideation, mania or depression requiring antidepressant therapy, or which could make it unsafe for the patient to participate in the opinion of the primary investigators
5. History of significant, unstable heart disease, including myocardial infarction, unstable angina, cardiac failure, second or third degree heart block, uncontrolled hypertension, syncope
6. Known hypersensitivity to cannabinoids or sesame oil
7. Any serious medical illness, which may require hospitalization during the study (i.e. sickle cell anemia, rheumatoid arthritis)
8. Has any disease of the gastrointestinal system, liver or kidneys which could result in altered metabolism or excretion of the study medication (history of major gastrointestinal tract surgery, gastrectomy, gastrotomy, bowel resection, etc.) or history of chronic gastrointestinal disorders (ulcerative colitis, regional enteritis, or gastrointestinal bleeding)
9. Female subjects who are pregnant or lactating, or female subjects of child bearing potential who are not using acceptable methods of birth control. Acceptable methods of birth control include:

   Barrier (diaphragm or condom) with spermicide, Intrauterine device, Levonorgestrel implant, Medroxyprogesterone acetate contraceptive injection, Oral contraceptives.
10. Clinical laboratory tests (CBC, blood chemistries, urinalysis) outside normal limits that are clinically unacceptable to the principal investigators. On EKG, 1st degree heart block, sinus tachycardia, left axis deviation, and nonspecific ST or T wave changes are allowed. Liver function tests (LFT's) <5 times ULN without symptoms of liver disease are acceptable after thorough medical review.

Additional Neuroimaging Exclusion Criteria:

Subjects who are selected for the clinical trial based on above inclusion and exclusion criteria will be screened further with the following exclusion criteria for possible participation in the fMRI imaging session:

1. Participation in a clinical trial and receipt of investigational drug(s) other than this clinical trial during previous 60 days.
2. History of serious head trauma or injury causing loss of consciousness that lasted more than 3 minutes.
3. Presence of magnetically active prosthetics, plates, pins, broken needles, permanent retainer, bullets, etc. in subject's body (unless a radiologist confirms that its presence is unproblematic). An X-ray may be obtained to determine eligibility.
4. Claustrophobia or other medical condition disabling subject from laying in the MRI for approximately 60 minutes

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2006-08; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles O'Brien, M.D./Ph.D., Principal Investigator — Treatment Research Center at the University of Pennsylvania
Locations (1):
- Treatment Research Center at the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Haney M, Hart CL, Vosburg SK, Nasser J, Bennett A, Zubaran C, Foltin RW. Marijuana withdrawal in humans: effects of oral THC or divalproex. Neuropsychopharmacology. 2004 Jan;29(1):158-70. doi: 10.1038/sj.npp.1300310. PMID 14560320
- [Derived] Goldman M, Szucs-Reed RP, Jagannathan K, Ehrman RN, Wang Z, Li Y, Suh JJ, Kampman K, O'Brien CP, Childress AR, Franklin TR. Reward-related brain response and craving correlates of marijuana cue exposure: a preliminary study in treatment-seeking marijuana-dependent subjects. J Addict Med. 2013 Jan-Feb;7(1):8-16. doi: 10.1097/ADM.0b013e318273863a. PMID 23188041

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All recruitment was conducted in West Philadelphia, PA, at the University of Pennsylvania Treatment Research Center, a facility providing treatment to study participants, between the years of 2007 and 2009.
Pre-assignment Details: All participants were screened with a number of medical and psychiatric evaluations prior to randomization to determine if they met study criteria.
Groups:
- All Screened Participants: All participants who met preliminary criteria and consented to undergo medical and psychiatric screening to determine eligibility for study randomization.
- Placebo 10mg QID; Dronabinol 10mg QID: All participants who were eligible for randomization, were randomized to receive either the active drug, dronabinol 10mg per dose up to 4 times per day or placebo up to 4 times per day.
Period: Screening
Arm/Group | All Screened Participants | Placebo 10mg QID | Dronabinol 10mg QID
Started | 61 | 0 (Participants did not enter this arm until period 3 "randomization") | 0 (Participants did not enter this arm until period 3 "randomization")
Completed | 24 | 0 (Participants did not enter this arm until period 3 "randomization") | 0 (Participants did not enter this arm until period 3 "randomization")
Not Completed | 37 | 0 | 0
Not completed — Not Eligible | 37 | 0 | 0
Period: Baseline Functional MRI
Arm/Group | All Screened Participants | Placebo 10mg QID | Dronabinol 10mg QID
Started | 24 (All non-randomized participants who also met specific eligibility for baseline functional MRI) | 0 (Participants did not enter this arm until period 3 "randomization") | 0 (Participants did not enter this arm until period 3 "randomization")
Completed | 12 | 0 (Participants did not enter this arm until period 3 "randomization") | 0 (Participants did not enter this arm until period 3 "randomization")
Not Completed | 12 | 0 | 0
Not completed — Functional MRI data not usable | 4 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0
Not completed — physical contraindication | 4 | 0 | 0
Period: Randomization
Arm/Group | All Screened Participants | Placebo 10mg QID | Dronabinol 10mg QID
Started | 0 | 13 | 11
Completed | 0 | 6 | 9
Not Completed | 0 | 7 | 2
Not completed — Lost to Follow-up | 0 | 7 | 2

BASELINE CHARACTERISTICS:
Population: 37 consented subjects were determined to be ineligible for randomization. This arm represents participants who were either given the placebo or dronabinol following the neuroimaging procedure.
  The only data available (summary level) is presented. Despite multiple good faith efforts, no access to individual data is available.
Groups:
- Non-Randomized Participants: These were participants who consented but were excluded prior to neuroimaging and randomization because they did not meet study criteria.
- Placebo/Dronabinol: This arm represents participants who were either given the placebo or dronabinol following the neuroimaging procedure. There was insufficient data to analyze the dronabinol and placebo groups separately due to an inability to meet statistical power considerations. Thus, for the results, the placebo and dronabinol subjects were combined into one group.
- Total: Total of all reporting groups
Arm/Group | Non-Randomized Participants | Placebo/Dronabinol | Total
Number analyzed (Participants) | 37 | 24 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.0 (10.4) | 37.6 (10.7) | 38.0 (10.4)
Sex/Gender, Customized [Number; unit: participants]
  Female | 8 | 5 | 13
  Male | 28 | 19 | 47
  Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 37 | 24 | 61

OUTCOME MEASURES:

1. Primary Outcome: Physiological Changes in Response to Cue-induced Craving.
Description: Functional MRI brain response to cannabis vs neutral cues. Higher T values represent increased blood flow in response to cues.
Time Frame: Baseline functional mri (fMRI), (prior to randomization)
Population: All participants who met preliminary criteria and consented to undergo medical and psychiatric screening to determine eligibility for study randomization.
Measure: Number; unit: T value
Groups:
- All Participants: All participants who met preliminary criteria and consented to undergo medical and psychiatric screening to determine eligibility for study randomization.
Arm/Group | All Participants
Number analyzed (Participants) | 12
T value | 5.65

2. Primary Outcome: Tolerability of Treatment
Description: Reports of side effects leading to discontinuation of treatment were examined in all participants.
Time Frame: baseline to two years
Population: Non-Randomized participants were not measured because they were not included in the neuroimaging study.
  The only data available (summary level) is presented. Despite all good faith efforts, no access to individual data is available.
Measure: Number; unit: participants
Groups:
- Placebo/Dronabinol: This arm represents the participants who, following neuroimaging procedure and randomization, were given either placebo or Dronabinol
Arm/Group | Non-Randomized Participants | Placebo/Dronabinol
Number analyzed (Participants) | 0 | 24
participants |  | 0

ADVERSE EVENTS:
Time Frame: two years
Description: Data was not collected separately for the Placebo and Dronabinol groups, but rather collected as a combined group.
Groups:
- Non-Randomized Participants: 37 consented subjects were determined to be ineligible for randomization.
- Placebo/Dronabinol: This arm represents participants who were either given the placebo or dronabinol following the neuroimaging procedure.
Arm/Group | Non-Randomized Participants | Placebo/Dronabinol
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/24
Other Adverse Events (participants affected / at risk) | 0/37 | 20/24
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-Randomized Participants (N=37) | Placebo/Dronabinol (N=24)
Change in Blood Pressure (Cardiac disorders) | 0 (0) | 2 (2)
Constipation/Diarrhea/ (Gastrointestinal disorders) | 0 (0) | 2 (2)
Loss of Appetite (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Cold/Flu Like (Infections and infestations) | 0 (0) | 4 (4)
Sedation/Drowsiness (Nervous system disorders) | 0 (0) | 9 (9)
Headache (Nervous system disorders) | 0 (0) | 4 (4)
Dysaesthesia (Nervous system disorders) | 0 (0) | 4 (4)
Depressed Mood (Psychiatric disorders) | 0 (0) | 1 (1)
High Feeling/Euphoria (Psychiatric disorders) | 0 (0) | 2 (2)
Increased Craving (Psychiatric disorders) | 0 (0) | 6 (6)
Irritable (Psychiatric disorders) | 0 (0) | 1 (1)
Createnine Elevation (mild) (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes